CLINICAL TRIAL: NCT06825741
Title: Brain Structural Abnormalities in Patients with Post-COVID-19 Headache
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: IG/296-1/2025/1
Record Dates: First submitted 2025-02-11; First posted 2025-02-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; Headache; MRI
Keywords: COVID-19; headache; MRI; brain; white matter lesion
MeSH Terms: conditions — COVID-19; Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Post-COVID-19 Headache Group: Participants in this group had a history of COVID-19 infection and developed persistent headaches afterward. They underwent brain MRI to assess potential structural abnormalities. Exclusion criteria included pre-existing neurological disorders or other conditions that could explain the headaches.
  Interventions: Other: Observational Study - No intervention
- Control Group: Participants in this group had no history of COVID-19 infection and no reported chronic headaches or neurological conditions. They underwent brain MRI for unrelated medical reasons and served as a comparison group to evaluate the prevalence of structural brain abnormalities in post-COVID headache patients.
  Interventions: Other: Observational Study - No intervention

INTERVENTIONS:
Other: Observational Study - No intervention — This is an observational study evaluating brain structural abnormalities in post-COVID headache patients. No experimental intervention is applied.

SUMMARY:
Introduction: The clinical manifestations of the COVID-19 pandemic are heterogeneous and may include various symptoms (gastrointestinal, musculoskeletal, neurological). Approximately 25% of patients report headache as a neurological symptom, making it the fifth most common symptom. These headaches may arise from structural brain changes associated with the infection.

Purpose: This study aims to identify the structural abnormalities observed in brain MRI that correlate with chronic headaches in patients who had COVID-19 infection.

Methods: The study included 30 patients with post-COVID-19 headaches and 30 control patients with no history of COVID-19. Demographic characteristics were analyzed using t-tests and chi-square tests. MRI findings were categorized into six types: cortical atrophy, white matter lesions, vascular lesions, lacunar lesions, vascular encephalopathy, and sinusitis. Differences in MRI findings between the two groups were evaluated using chi-square tests. Secondary outcomes included the analysis of symptoms accompanying headaches, diagnoses following MRI, and treatments applied.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of COVID-19 infection
* Persistent headache following COVID-19 infection
* Brain MRI requested by the attending physician

Exclusion Criteria:

* Prior neurological disease or disorder
* MRI contraindications (e.g., pacemaker, metal implants, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients (≥18 years) with persistent headaches following COVID-19 infection who were referred for brain MRI to investigate potential structural abnormalities. A control group of individuals without a history of COVID-19 infection or chronic headaches was included for comparison. Exclusion criteria included prior neurological diseases, recent head trauma, and MRI contraindications.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Specific Structural Brain Abnormalities Observed on MRI | From September 2020 to December 2022
  Brain MRI scans were analyzed to determine the number of participants with specific structural abnormalities, including white matter lesions, cortical atrophy, vascular encephalopathy, lacunar infarcts, and sinusitis. Each abnormality was evaluated separately, and the number of participants affected by each type was recorded.

SECONDARY OUTCOMES:
Number of Participants Reporting Additional Symptoms Associated with Post-COVID-19 Headache | From September 2020 to December 2022
  The number of participants experiencing symptoms such as dizziness, cognitive dysfunction, and visual disturbances was recorded. Each symptom was assessed separately and reported as the number of affected participants.
Number of Participants Diagnosed with Specific Conditions After MRI | From September 2020 to December 2022
  Following MRI evaluation, the number of participants diagnosed with specific conditions (e.g., migraines, post-COVID headache, vestibular syndrome) was recorded. Each diagnosis was evaluated and reported separately.
Number of Participants Receiving Specific Treatment Approaches for Post-COVID-19 Headache | From September 2020 to December 2022
  The number of participants receiving pharmacological treatments (e.g., cognitive enhancers, antidepressants) and lifestyle modifications was recorded. Each treatment approach was assessed separately and reported as the number of affected participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Szent Margit Hospital, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Szephelyi K, Kora S, Orsi G, Tollar J. Brain Structural Abnormalities in Patients with Post-COVID-19 Headache. Neurol Int. 2025 Mar 26;17(4):50. doi: 10.3390/neurolint17040050. PMID 40278421